CLINICAL TRIAL: NCT04025684
Title: Randomized Controlled Examiner-Blind Methodology Development Study To Investigate The Plaque Removal Efficacy Of Manual Toothbrushes In Healthy Dentate Subjects
Brief Title: Efficacy of Manual Toothbrushes in Removing Dental Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 212224
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Dental Plaque; Oral Hygiene
Keywords: Oral Hygiene
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Examiner-blind; Monitor and Data-analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test toothbrush 1 (Other): Participants will brush their entire dentition twice daily (morning and evening) for 1-timed minute with test toothbrush 1 after applying a strip of standard fluoride (1450 parts per million [ppm] fluoride) toothpaste (full brush head) and will then rinse with 10 mL of water post brushing for 5 seconds (on site). Offsite participants will be permitted to rinse with tap water according to their normal habitat.
  Interventions: Other: Oral B Indicator 123
- Test toothbrush 2 (Other): Participants will brush their entire dentition twice daily (morning and evening) for 1-timed minute with test toothbrush 2 after applying a strip of standard fluoride (1450 ppm fluoride) toothpaste (full brush head) and will then rinse with 10 mL of water post brushing for 5 seconds (on site). Offsite participants will be permitted to rinse with tap water according to their normal habitat.
  Interventions: Other: Dr Best Original
- Test toothbrush 3 (Other): Participants will brush their entire dentition twice daily (morning and evening) for 1-timed minute with test toothbrush 3 after applying a strip of standard fluoride (1450 ppm fluoride) toothpaste (full brush head) and will then rinse with 10 mL of water post brushing for 5 seconds (on site). Offsite participants will be permitted to rinse with tap water according to their normal habitat.
  Interventions: Other: Dr Best Multi Expert
- Test toothbrush 4 (Other): Participants will brush their entire dentition twice daily (morning and evening) for 1-timed minute with test toothbrush 4 after applying a strip of standard fluoride (1450 ppm fluoride) toothpaste (full brush head) and will then rinse with 10 mL of water post brushing for 5 seconds (on site). Offsite participants will be permitted to rinse with tap water according to their normal habitat.
  Interventions: Other: parodontax Interdental

INTERVENTIONS:
Other: Oral B Indicator 123 — Manual toothbrush (medium bristle stiffness; compact head, UK market).
  Arms: Test toothbrush 1
Other: Dr Best Original — Manual toothbrush (medium bristle stiffness; regular head, German market)
  Arms: Test toothbrush 2
Other: Dr Best Multi Expert — Manual toothbrush (medium bristle stiffness; compact head, German market)
  Arms: Test toothbrush 3
Other: parodontax Interdental — Manual toothbrush (soft bristle stiffness; compact head, German market)
  Arms: Test toothbrush 4

SUMMARY:
This clinical methodology development study will evaluate the plaque removal efficacy of four marketed manual toothbrushes, with differing bristle types and brush head designs, in healthy dentate participants. Changes in supra-gingival plaque accumulation will be assessed after first use and following 1-and 4-weeks treatment (twice-daily brushing), using two different clinical measures of dental plaque. Study participants will abstain from oral hygiene for a period of 12-18 hours prior to each assessment visit. Data generated will inform the design of future clinical studies investigating the plaque removal efficacy of manual toothbrushes.

DETAILED DESCRIPTION:
This will be a single center, 4-week, randomized, controlled, examiner-blind, four-treatment arm, parallel design, clinical methodology development study to investigate the plaque removal efficacy of marketed manual toothbrushes in healthy, dentate participants. Changes in plaque level will be evaluated after first brushing, after two further single brushing events (Days 7 and 28) and following 7 and 28 days usage (twice daily brushing with assigned toothbrush treatment).

Supra-gingival plaque levels will be assessed using two established clinical measures: the Rustogi Modified Navy Plaque Index (RPI) and the 6-site Turesky Modified Quigley and Hein Plaque Index (TPI). Participants will abstain from oral hygiene for a period of 12-18 hours prior to each assessment visit. Participants with Day 0 pre-brushing mean RPI overall ≥ 0.6 will be stratified by their Day 0 pre-brushing RPI score (lower: mean RPI overall ≥ 0.6 to ≤ 0.8; higher: mean RPI overall; 0.8 to 1.0) and randomized to study treatment (Visit 2).

To standardize oral hygiene practice, eligible participants will complete a lead-in period (minimum 5 days) prior to Visit 2 during which they will brush with the toothbrush and regular fluoride toothpaste provided.

The safety and oral tolerability of each study toothbrush will be monitored after first use and over the 28-day usage period by review of reported treatment emergent adverse events (TEAEs).

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all the following inclusion criteria to be eligible for enrollment into the study.

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant in good general, mental and oral health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, well-being or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant with, in the opinion of the investigator or medically qualified designee, satisfactory oral hygiene based on oral examination.
* A participant who routinely uses a manual toothbrush for daily oral hygiene.
* VISIT 1 (Screening): A participant must have a) ≥ 20 natural, permanent teeth b) ≥ 40 gradable tooth surfaces (≥ 2/3rds of the tooth surface assessable for RPI).Third molars, fully crowned/ extensively restored, grossly carious, orthodontically-banded/bonded or abutment teeth and surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with plaque assessment should not be included in the gradable surface count. Third molars can be included if, as a result tooth loss, they are functioning as second molars.
* VISIT 2 (Baseline): A participant must have a pre-brushing mean RPI ≥ 0.6 overall (that is, the mean over all gradable surfaces)

Exclusion Criteria:

An individual who meets any of the following exclusion criteria will not be eligible for enrollment into the study.

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or otherwise supervised by the investigator, or a member of their immediate family; or a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) in the 30 days prior to study entry and/or who is participating in other studies during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant with any medical/oral condition which, in the opinion of the investigator or medically qualified designee, could impact study outcomes (for example, oral dryness).
* A participant taking daily doses of medication/having daily treatments which, in the opinion of the investigator or medically qualified designee, could impact study outcomes (for example, is causing oral dryness).
* A participant with any condition or physical limitation which, in the opinion of the investigator or medically qualified designee, impacts their ability to perform oral hygiene with a manual toothbrush.
* A participant who is pregnant (self-reported; no pregnancy test required) or intending to become pregnant over the course of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who is unwilling or unable to comply with the following Lifestyle Considerations described in this protocol: 1) Dental Product/Treatment and Oral Hygiene Restrictions i)From Screening (Visit 1) to the Participant's Last Study Visit: a) Participants should not use any other oral care products (for example, toothpastes, toothbrushes, oral rinses, tongue cleaners, whitening/bleaching products, inter-dental cleaning products)than those provided during the study. Note: dental floss (non-antibacterial) can be used to remove impacted food; b) Participants should not chew gum or consume any confectionery containing xylitol (e.g. sugar-free mints); c) Participants should delay any non-emergency dental treatment until after study completion (including dental prophylaxis); d)Participants should delay any tooth whitening treatments (professional and/or home use) until after study completion; ii) Before Clinical Efficacy Assessment Visits (Visits 2-4): Participants should refrain from oral hygiene procedures for 12-18 hours before their visit; 2) Meals and Dietary Restrictions i) Before Clinical Efficacy Assessment Visits (Visits 2-4): Participants should not eat or drink for ≥ 1 hour before their visit and until all visit procedures have been completed.
* A participant who has had routine dental prophylaxis within 4 weeks of Screening.
* A participant who has undergone a tooth bleaching procedure within 8 weeks of Screening.
* A participant with, in the opinion of the investigator or medically qualified designee, generalized moderate/severe gingivitis.
* A participant with, in the opinion of the investigator or medically qualified designee, gross periodontal disease.
* A participant with, in the opinion of the investigator or medically qualified designee, signs of active periodontitis.
* A participant with a Basic Periodontal Examination (BPE) score ≥ 3 in any sextant.
* A participant who has undergone treatment for periodontal disease within 12 months of Screening, including scaling and/or root surface debridement.
* A participant who is currently undergoing treatment for periodontal disease, including scaling and/or root surface debridement.
* A participant with active caries which, in the opinion of the investigator or medically qualified designee, could impact study outcomes or the oral health of the participant if they were to participate in the study.
* A participant with, in the opinion of the investigator or medically qualified designee, evidence of gross intra-oral neglect or the need for extensive dental therapy.
* A participant with restorations in a poor state of repair which, in the opinion of the investigator or medically qualified designee, could impact study outcomes.
* A participant with any dental condition (e.g. malalignment, overcrowding) which, in the opinion of the investigator or medically qualified designee, could impact study outcomes.
* A participant with high levels of extrinsic dental stain or calculus deposits which, in the opinion of the investigator or medically qualified designee, would interfere with plaque assessment or impact study outcomes.
* A participant with a tongue or lip piercing.
* A participant with multiple dental implants which, in the opinion of the investigator or medically qualified designee, could impact study outcomes.
* A participant with fixed bridge(s) or removable partial dentures.
* A participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* A participant who has had fixed or removable orthodontic braces/bands within 3 months of Screening.
* A participant who is unwilling to forgo use of an orthodontic retainer for the duration of the study, provided there would be no impact on the outcome of any previous, completed orthodontic treatment or the participant's well-being.
* VISIT 1 (Screening): A participant who has taken antibiotics within 2 weeks of Screening.
* VISIT 2 (Baseline): A participant who has taken antibiotics during the lead-in period (between Screening and Visit 2).
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of primary endpoints of the study.
Access Criteria: Access is provided after a research proposal submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United Kingdom.
Pre-assignment Details: A total of 125 participants were screened, of whom 80 were randomized in 4 study product groups, 33 did not meet the study criteria, 2 were lost to follow-up, 2 withdrew consent, and 8 were not randomized due to other reason.
Groups:
- Oral B Indicator 123: Participants randomized to this group dosed the Oral B Indicator 123 toothbrush with a strip of regular fluoride toothpaste (full brush head) and then brushed their entire dentition for 1 timed minute, twice daily (morning and evening) and rinsed with 10 milliliters (mL) tap water post-brushing for 5 seconds while brushing on-site and with tap water post-brushing, according to their normal habit while brushing off-site. Overall study duration was 30 days.
- Dr Best Original: Participants randomized to this group dosed the Dr Best Original toothbrush with a strip of regular fluoride toothpaste (full brush head) and then brushed their entire dentition for 1 timed minute, twice daily (morning and evening) and rinsed with 10 mL tap water post-brushing for 5 seconds while brushing on-site and with tap water post-brushing, according to their normal habit while brushing off-site. Overall study duration was 30 days.
- Dr Best Multi Expert: Participants randomized to this group dosed the Dr Best Multi Expert toothbrush with a strip of regular fluoride toothpaste (full brush head) and then brushed their entire dentition for 1 timed minute, twice daily (morning and evening) and rinsed with 10 mL tap water post-brushing for 5 seconds while brushing on-site and with tap water post-brushing, according to their normal habit while brushing off-site. Overall study duration was 30 days.
- Parodontax Interdental: Participants randomized to this group dosed the parodontax Interdental toothbrush with a strip of regular fluoride toothpaste (full brush head) and then brushed their entire dentition for 1 timed minute, twice daily (morning and evening) and rinsed with 10 mL tap water post-brushing for 5 seconds while brushing on-site and with tap water post-brushing, according to their normal habit while brushing off-site. Overall study duration was 30 days.
Period: Overall Study
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Started | 20 | 19 | 20 | 21
Completed | 18 | 15 | 20 | 20
Not Completed | 2 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Multiple reasons | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who completed at least one use of study product.
Groups:
- Oral B Indicator 123: Participants randomized to this group dosed the Oral B Indicator 123 toothbrush with a strip of regular fluoride toothpaste (full brush head) and then brushed their entire dentition for 1 timed minute, twice daily (morning and evening) and rinsed with 10 mL tap water post-brushing for 5 seconds while brushing on-site and with tap water post-brushing, according to their normal habit while brushing off-site. Overall study duration was 30 days.
- Total: Total of all reporting groups
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental | Total
Number analyzed (Participants) | 20 | 19 | 20 | 21 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 20 | 20 | 79
  >=65 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 10 | 16 | 52
  Male | 6 | 7 | 10 | 5 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 1 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 4 | 1 | 9
  White | 12 | 16 | 15 | 19 | 62
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre to Post Brushing in Overall Mean Rustogi Modified Navy Plaque Index (RPI) After a Single Brushing Event at Day 0
Description: Supra-gingival plaque was assessed on the facial and lingual surfaces of the teeth (7-7 each arch) using RPI. Each tooth surface was divided into 9 zones, for a total of 18 sites per tooth (A to I facial with 9 sites and lingual with 9 sites separately); A to C along gingival margin; D to F directly above A to C (D and F being inter-proximal zones); G to H across middle of tooth; and I covered incisal area. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from pre-brushing = (post-brushing score - pre-brushing score). Overall mean calculated for all participants was reported.
Time Frame: At Day 0
Population: Modified intent-to-treat population (mITT) comprised all randomized participants who had a postbaseline plaque assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale | -0.09623 (0.052741) | -0.12005 (0.055350) | -0.09859 (0.045509) | -0.09599 (0.044436)
Statistical Analysis 1: Comparison: Oral B Indicator 123; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < .0001, ANCOVA — Analysis was performed using ANCOVA Model with product group as a fixed effect and the baseline mean RPI overall value as a covariate; Adjusted Mean Change = -0.10, 95% CI 2-sided [-0.11 to -0.08], Standard Error of Mean 0.010
Statistical Analysis 2: Comparison: Dr Best Original; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Change = -0.12, 95% CI 2-sided [-0.14 to -0.10], Standard Error of Mean 0.010
Statistical Analysis 3: Comparison: Dr Best Multi Expert; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Change = -0.10, 95% CI 2-sided [-0.12 to -0.08], Standard Error of Mean 0.010
Statistical Analysis 4: Comparison: Parodontax Interdental; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Change = -0.10, 95% CI 2-sided [-0.12 to -0.08], Standard Error of Mean 0.010

2. Primary Outcome: Change From Pre to Post Brushing in Overall Mean Turesky Modified Quigley & Hein Plaque Index (TPI) After a Single Brushing Event at Day 0
Description: Supra-gingival plaque accumulation was assessed on facial and lingual surfaces of teeth (7-7 in each arch) using TPI. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1millimetre [mm] or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from pre-brushing = (post-brushing score - pre-brushing score). Overall mean calculated for all participants was reported.
Time Frame: At Day 0
Population: mITT comprised all randomized participants who had a postbaseline plaque assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
Score on a scale | -0.49354 (0.312963) | -0.62218 (0.340491) | -0.57721 (0.347314) | -0.53714 (0.273720)
Statistical Analysis 1: Comparison: Oral B Indicator 123; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — Analysis was performed using ANCOVA model with product group as a fixed effect, and the baseline mean TPI overall value and RPI stratification level as covariates; Adjusted Mean Change = -0.50, 95% CI 2-sided [-0.62 to -0.37], Standard Error of Mean 0.065
Statistical Analysis 2: Comparison: Dr Best Original; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted Mean Change = -0.62, 95% CI 2-sided [-0.75 to -0.49], Standard Error of Mean 0.066
Statistical Analysis 3: Comparison: Dr Best Multi Expert; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted Mean Change = -0.55, 95% CI 2-sided [-0.68 to -0.42], Standard Error of Mean 0.066
Statistical Analysis 4: Comparison: Parodontax Interdental; Statistical analysis was performed with comparison in pre-treatment and post-treatment within the treatment group; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted Mean Change = -0.57, 95% CI 2-sided [-0.70 to -0.44], Standard Error of Mean 0.066

3. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) to Post-Brushing in Overall Mean Rustogi Modified Navy Plaque Index (RPI) at Day 7 and Day 28
Description: Supra-gingival plaque was assessed on the facial and lingual surfaces of the teeth (7-7 each arch) using RPI. Each tooth surface was divided into 9 zones, for a total of 18 sites per tooth (A to I facial with 9 sites and lingual with 9 sites separately); A to C along gingival margin; D to F directly above A to C (D and F being inter-proximal zones); G to H across middle of tooth; and I covered incisal area. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28 = (post-brushing score at Day 7/28- pre-brushing score at Day 0). Overall mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: mITT comprised all randomized participants who had a postbaseline plaque assessment. Here, number analyzed indicates participants with available data for each category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Change at Day 7 Post brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  Change at Day 7 Post brushing | -0.13485 (0.057076) | -0.16648 (0.074227) | -0.09813 (0.068715) | -0.11839 (0.059674)
  Change at Day 28 Post brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  Change at Day 28 Post brushing | -0.14738 (0.071082) | -0.16234 (0.047753) | -0.12854 (0.085085) | -0.11835 (0.070860)

4. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) to Post-Brushing in Overall Mean Turesky Modified Quigley & Hein Plaque Index (TPI) at Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed on facial and lingual surfaces of teeth (7-7 in each arch) using TPI. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1mm or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28 = (post-brushing score at Day 7/28- pre-brushing score at Day 0). Overall mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Change at Day 7 Post brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  Change at Day 7 Post brushing | -0.71646 (0.290669) | -0.90569 (0.436986) | -0.63582 (0.417132) | -0.61935 (0.348844)
  Change at Day 28 Post brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  Change at Day 28 Post brushing | -0.75755 (0.330047) | -0.79959 (0.281520) | -0.70769 (0.438260) | -0.60327 (0.379847)

5. Secondary Outcome: Overall Mean Rustogi Modified Navy Plaque Index (RPI) Pre- and Post-brushing at Day 7 and Day 28
Description: Supra-gingival plaque was assessed on the facial and lingual surfaces of the teeth (7-7 each arch) using RPI. Each tooth surface was divided into 9 zones, for a total of 18 sites per tooth (A to I facial with 9 sites and lingual with 9 sites separately); A to C along gingival margin; D to F directly above A to C (D and F being inter-proximal zones); G to H across middle of tooth; and I covered incisal area. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Overall mean calculated for all participants was reported.
Time Frame: At Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 7 Pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Pre-brushing | 0.443 (0.0739) | 0.438 (0.0859) | 0.468 (0.0738) | 0.449 (0.0654)
  At Day 7 Post-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Post-brushing | 0.352 (0.0695) | 0.333 (0.0749) | 0.390 (0.0924) | 0.352 (0.0681)
  At Day 28 Pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Pre-brushing | 0.443 (0.0920) | 0.467 (0.0888) | 0.467 (0.0721) | 0.434 (0.0756)
  At Day 28 Post-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Post-brushing | 0.340 (0.1113) | 0.343 (0.0974) | 0.360 (0.0802) | 0.352 (0.0736)

6. Secondary Outcome: Overall Mean Turesky Modified Quigley & Hein Plaque Index (TPI) Pre- and Post-brushing TPI at Day 7, and Day 28
Description: Supra-gingival plaque accumulation was assessed on facial and lingual surfaces of teeth (7-7 in each arch) using TPI. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1mm or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Overall mean calculated for all participants was reported.
Time Frame: At Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 7 Pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Pre-brushing | 2.361 (0.4198) | 2.368 (0.5218) | 2.508 (0.4270) | 2.446 (0.3834)
  At Day 7 Post-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Post-brushing | 1.803 (0.4084) | 1.669 (0.4246) | 1.945 (0.5175) | 1.816 (0.3902)
  At Day 28 Pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Pre-brushing | 2.327 (0.5263) | 2.459 (0.4062) | 2.452 (0.2773) | 2.346 (0.3421)
  At Day 28 Post-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Post-brushing | 1.766 (0.5549) | 1.788 (0.5161) | 1.870 (0.4209) | 1.832 (0.4330)

7. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) to Post-Brushing in Gingival Margin Sites Mean Rustogi Modified Navy Plaque Index (RPI) at Day 0, Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed for gingival zone A to C. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 0/7/28= (post-brushing score at Day 0/7/28- pre-brushing score at Day 0). Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Change at Day 0 Post brushing | -0.04938 (0.054115) | -0.09034 (0.092453) | -0.05344 (0.059657) | -0.07211 (0.058880)
  Change at Day 7 Post brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  Change at Day 7 Post brushing | -0.12498 (0.096075) | -0.16961 (0.132531) | -0.09456 (0.095039) | -0.12165 (0.089975)
  Change at Day 28 Post brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  Change at Day 28 Post brushing | -0.17348 (0.152077) | -0.16314 (0.156324) | -0.12075 (0.123455) | -0.10500 (0.110297)

8. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) to Post-Brushing in Inter-Proximal Sites Mean Rustogi Modified Navy Plaque Index (RPI) at Day 0, Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed for inter-proximal zones D to F. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 0/7/28= (post-brushing score at Day 0/7/28- pre-brushing score at Day 0). Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Change at Day 0 Post brushing | -0.26809 (0.130993) | -0.28219 (0.133379) | -0.25775 (0.123545) | -0.22865 (0.130830)
  Change at Day 7 Post brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  Change at Day 7 Post brushing | -0.31485 (0.161214) | -0.33171 (0.188937) | -0.21269 (0.167972) | -0.24499 (0.172251)
  Change at Day 28 Post brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  Change at Day 28 Post brushing | -0.30399 (0.153080) | -0.32138 (0.130552) | -0.26825 (0.188777) | -0.25411 (0.191171)

9. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) to Post-Brushing in Inter-Proximal Sites Mean Turesky Modified Quigley & Hein Plaque Index (TPI) at Day 0, Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed for inter-proximal zones D to F. Plaque was disclosed and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1mm or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 0/7/28= (post-brushing score at Day 0/7/28- pre-brushing score at Day 0). Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Change at Day 0 Post brushing | -0.49949 (0.314629) | -0.60975 (0.337375) | -0.58666 (0.352225) | -0.49861 (0.291868)
  Change at Day 7 Post brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  Change at Day 7 Post brushing | -0.72054 (0.293855) | -0.89035 (0.429582) | -0.62843 (0.400444) | -0.56209 (0.365074)
  Change at Day 28 Post brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  Change at Day 28 Post brushing | -0.78797 (0.326878) | -0.81581 (0.261399) | -0.72924 (0.445553) | -0.58135 (0.389490)

10. Secondary Outcome: Gingival Margin Sites Mean Rustogi Modified Navy Plaque Index (RPI) Pre- and Post-brushing at Day 0, Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed for gingival zone A to C. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 0 Pre-brushing | 0.988 (0.0227) | 0.987 (0.0213) | 0.992 (0.0115) | 0.981 (0.0481)
  At Day 0 Post-brushing | 0.939 (0.0635) | 0.896 (0.0932) | 0.939 (0.0577) | 0.909 (0.0894)
  At Day 7 Pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Pre-brushing | 0.966 (0.0488) | 0.952 (0.0831) | 0.978 (0.0376) | 0.969 (0.0406)
  At Day 7 Post-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Post-brushing | 0.863 (0.1046) | 0.818 (0.1429) | 0.898 (0.0931) | 0.859 (0.1056)
  At Day 28 Pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Pre-brushing | 0.945 (0.1094) | 0.974 (0.0436) | 0.983 (0.0252) | 0.964 (0.0657)
  At Day 28 Post-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Post-brushing | 0.814 (0.1625) | 0.825 (0.1686) | 0.871 (0.1218) | 0.876 (0.1127)

11. Secondary Outcome: Inter-Proximal Sites Mean Rustogi Modified Navy Plaque Index (RPI) Pre- and Post-brushing at Day 0, Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed for inter-proximal zones D to F. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 0 Pre-brushing | 0.523 (0.2121) | 0.499 (0.2217) | 0.507 (0.1626) | 0.467 (0.1910)
  At Day 0 Post-brushing | 0.255 (0.1551) | 0.217 (0.1611) | 0.249 (0.1422) | 0.238 (0.1397)
  At Day 7 Pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Pre-brushing | 0.389 (0.2041) | 0.371 (0.2083) | 0.453 (0.1969) | 0.408 (0.1668)
  At Day 7 Post-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Post-brushing | 0.214 (0.1344) | 0.191 (0.1080) | 0.294 (0.2048) | 0.222 (0.1187)
  At Day 28 Pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Pre-brushing | 0.431 (0.2299) | 0.442 (0.2341) | 0.479 (0.2370) | 0.381 (0.2083)
  At Day 28 Post-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Post-brushing | 0.227 (0.2136) | 0.217 (0.1478) | 0.239 (0.1666) | 0.213 (0.1640)

12. Secondary Outcome: Inter-Proximal Sites Mean Turesky Modified Quigley & Hein Plaque Index (TPI) Pre- and Post-brushing TPI at Day 0, Day 7 and Day 28
Description: Supra-gingival plaque accumulation was assessed for inter-proximal zones D to F. Plaque was disclosed and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1mm or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 0 Pre-brushing | 2.643 (0.3965) | 2.649 (0.4338) | 2.737 (0.3425) | 2.552 (0.4292)
  At Day 0 Post-brushing | 2.141 (0.3735) | 2.041 (0.3815) | 2.149 (0.2642) | 2.054 (0.4217)
  At Day 7 Pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Pre-brushing | 2.481 (0.4396) | 2.493 (0.4949) | 2.635 (0.4564) | 2.577 (0.4149)
  At Day 7 Post-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Post-brushing | 1.937 (0.4208) | 1.821 (0.4075) | 2.109 (0.5191) | 1.991 (0.3755)
  At Day 28 Pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Pre-brushing | 2.410 (0.5228) | 2.550 (0.3968) | 2.561 (0.2938) | 2.454 (0.3358)
  At Day 28 Post-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Post-brushing | 1.871 (0.5645) | 1.911 (0.4994) | 2.007 (0.4122) | 1.972 (0.4141)

13. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) in Overall Rustogi Modified Navy Plaque Index (RPI) at Day 7 Pre-brushing and Day 28 Pre-brushing
Description: Supra-gingival plaque was assessed on the facial and lingual surfaces of the teeth (7-7 each arch) using RPI. Each tooth surface was divided into 9 zones, for a total of 18 sites per tooth (A to I facial with 9 sites and lingual with 9 sites separately); A to C along gingival margin; D to F directly above A to C (D and F being inter-proximal zones); G to H across middle of tooth; and I covered incisal area. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28= (pre-brushing score at Day 7/28- pre-brushing score at Day 0). Overall mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 pre-brushing and Day 28 pre-brushing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 7 Pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 Pre-brushing | -0.04465 (0.060772) | -0.06178 (0.058426) | -0.01992 (0.050254) | -0.02163 (0.056758)
  At Day 28 Pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 Pre-brushing | -0.04420 (0.060384) | -0.03796 (0.060434) | -0.02121 (0.061780) | -0.03689 (0.075670)

14. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) in Overall Mean Turesky Modified Quigley & Hein Plaque Index (TPI) at Day 7 Pre-brushing and Day 28 Pre-brushing
Description: Supra-gingival plaque accumulation was assessed on facial and lingual surfaces of teeth (7-7 in each arch) using TPI. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1mm or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28= (pre-brushing score at Day 7/28- pre-brushing score at Day 0). Overall mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 pre-brushing and Day 28 pre-brushing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 7 pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 pre-brushing | -0.15663 (0.307019) | -0.20746 (0.360506) | -0.07029 (0.315099) | 0.01187 (0.282108)
  At Day 28 pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 pre-brushing | -0.19667 (0.343446) | -0.12896 (0.236209) | -0.12756 (0.302698) | -0.08991 (0.357293)

15. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) in Gingival Margin Sites Mean Rustogi Modified Navy Plaque Index (RPI) at Day 7 Pre-brushing and Day 28 Pre-brushing
Description: Supra-gingival plaque accumulation was assessed for gingival zone A to C. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28= (pre-brushing score at Day 7/28- pre-brushing score at Day 0). Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 pre-brushing and Day 28 pre-brushing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 7 pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 pre-brushing | -0.02233 (0.035312) | -0.03645 (0.066621) | -0.01378 (0.040284) | -0.01219 (0.038447)
  At Day 28 pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 pre-brushing | -0.04272 (0.100638) | -0.01355 (0.034877) | -0.00943 (0.026501) | -0.01715 (0.083641)

16. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) in Inter-Proximal Sites Mean Rustogi Modified Navy Plaque Index (RPI) at Day 7 Pre-brushing and Day 28 Pre-brushing
Description: Supra-gingival plaque accumulation was assessed for inter-proximal zones D to F. Plaque was disclosed and presence or absence of plaque in each zone was recorded as per scoring criteria: 0-Plaque absent, 1-Plaque present; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28= (pre-brushing score at Day 7/28- pre-brushing score at Day 0). Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 pre-brushing and Day 28 pre-brushing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  At Day 7 pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 pre-brushing | -0.13944 (0.184635) | -0.15199 (0.162624) | -0.05413 (0.144292) | -0.05919 (0.175623)
  At Day 28 pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 pre-brushing | -0.09970 (0.132324) | -0.09659 (0.197697) | -0.02755 (0.204586) | -0.08592 (0.215974)

17. Secondary Outcome: Change From Baseline (Day 0 Pre-Brushing) in Inter-Proximal Sites Mean Turesky Modified Quigley & Hein Plaque Index (TPI) at Day 7 Pre-brushing and Day 28 Pre-brushing
Description: Supra-gingival plaque accumulation was assessed for inter-proximal zones D to F. Plaque was disclosed and scored for each site on a scale of 0 to 5: 0-No plaque, 1-Slight flecks of plaque at cervical margin of tooth, 2-Thin, continuous band of plaque (1mm or smaller) at cervical margin of tooth, 3-Band of plaque wider than 1mm but covering less than 1/3 of area, 4-Plaque covering at least 1/3 but less than 2/3 of area, 5-Plaque covering 2/3 or more of crown of tooth; where lower score represents better result. An average score for a participant was generated by averaging across all sites and surfaces of all teeth assessed. Change from Day 0 pre-brushing at Day 7/28= (pre-brushing score at Day 7/28- pre-brushing score at Day 0). Mean calculated for all participants was reported.
Time Frame: At Day 0, Day 7 pre-brushing and Day 28 pre-brushing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
Number analyzed (Participants) | 20 | 19 | 20 | 20
Score on a scale
  At Day 7 pre-brushing: number analyzed (Participants) | 19 | 16 | 20 | 20
  At Day 7 pre-brushing | -0.17652 (0.309335) | -0.21666 (0.366396) | -0.10226 (0.315550) | 0.02326 (0.316914)
  At Day 28 pre-brushing: number analyzed (Participants) | 18 | 15 | 20 | 20
  At Day 28 pre-brushing | -0.25042 (0.332584) | -0.17761 (0.225399) | -0.17561 (0.327045) | -0.09889 (0.370219)

ADVERSE EVENTS:
Time Frame: Up to 35 days
Description: Safety population included all randomized participants who completed at least one use of study product. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported. A participant with multiple occurrences of AEs counted once in AE category. A participant with multiple AEs within a primary system organ class was counted once in system organ class.
Arm/Group | Oral B Indicator 123 | Dr Best Original | Dr Best Multi Expert | Parodontax Interdental
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 2/19 | 1/20 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral B Indicator 123 (N=20) | Dr Best Original (N=19) | Dr Best Multi Expert (N=20) | Parodontax Interdental (N=21)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04025684/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT04025684/SAP_001.pdf